CLINICAL TRIAL: NCT01506752
Title: A Bioequivalence Study Comparing Improved Versus Current Orally Disintegrating E2020 10 mg Tablet in Healthy Japanese Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: E2020-J081-034
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-01

CONDITIONS: Healthy Adult
Keywords: Bioequivalence; Healthy Subjects; Donepezil
MeSH Terms: interventions — Donepezil

ARMS (4):
- E2020 improved 10 mg without water (Active Comparator)
  Interventions: Drug: Donepezil Hydrochloride
- E2020 current 10 mg without water (Active Comparator)
  Interventions: Drug: Donepezil Hydrochloride
- E2020 improved 10 mg with water (Active Comparator)
  Interventions: Drug: Donepezil Hydrochloride
- E2020 current 10 mg with water (Active Comparator)
  Interventions: Drug: Donepezil Hydrochloride

INTERVENTIONS:
Drug: Donepezil Hydrochloride — improved orally disintegrating E2020 10 mg tablet without water.
  Arms: E2020 improved 10 mg without water
Drug: Donepezil Hydrochloride — current orally disintegrating E2020 10 mg tablet without water.
  Arms: E2020 current 10 mg without water
Drug: Donepezil Hydrochloride — improved orally disintegrating E2020 10 mg tablet with water.
  Arms: E2020 improved 10 mg with water
Drug: Donepezil Hydrochloride — current orally disintegrating E2020 10 mg tablet with water
  Arms: E2020 current 10 mg with water

SUMMARY:
The purpose of this study is to investigate the bioequivalence of improved and current orally disintegrating E2020 10 mg tablets as a single dose in Japanese healthy adult males for each of two administration methods (with/without water).

ELIGIBILITY:
Inclusion Criteria

Those who meet all below criteria are eligible to enroll in this study;

1. Those who provide consent by their own will.
2. Male subjects aged between ≥ 20 years and < 45 years old at the time of obtaining informed consent and non-smoker (subjects who have not been smoking for at least 4 weeks prior to study treatment)
3. BMI at screening is 18.5 kg/m2 or above and less than 25.0 kg/m2
4. Those who are willing to and can comply with the conditions described in the study protocol.

Exclusion Criteria

Those who meet any of the below criteria will be excluded from the study.

1. Any significant medical illness that required intervention within 8 weeks before treatment, or any medical history of clinically significant infectious diseases within 4 weeks before treatment.
2. Those who had any psychiatric, GI tract, hepatic, renal, respiratory, endocrine, hematological, neurological, cardiovascular diseases or congenital metabolic disorders within 4 weeks before study drug administration that may have an impact on the evaluation of the drug.
3. Subjects who have any medical history of GI, hepatic, or renal surgery (e.g. excision of liver, kidney or GI tract) that may have an impact on pharmacokinetics of the drug.
4. Subjects who have any history of medically significant allergy to medications or foods, and those who currently have any symptoms of seasonal
5. Subjects whose weight changes were more than 10% from the screening phase to study drug administration.
6. Those with clinical abnormal symptoms, medical history of organ dysfunction, subjective symptoms, objective findings, vital signs, and abnormal EKG or clinical laboratory test values, which need medical intervention.
7. Corrected change in QT wave (QTc) interval of > 450 msec with 12-lead EKG at screening or study drug administration.
8. Subjects who are positive for hepatitis B surface antigen (HBs antigen), hepatitis C (HCV) antibody, or serologic test for syphilis (STS).
9. Subjects who are suspected with or who has a history of drug or alcohol abuse, or positive urine screen for drugs of abuse or exhalation alcohol test at screening or baseline.
10. Subjects who consumed caffeine-containing food or beverages within 72 hours before study drug administration.
11. Exposure to any supplements or herbs (including Chinese medicine), or beverages (e.g. alcohol or grapefruit-containing beverages, within 2 weeks of study drug administration.
12. Exposure to St. John's wort containing medications within 4 weeks of study drug administration.
13. Use of any prescription drugs within 4 week before study drug administration.
14. Use of any OTC medications within 2 week before study drug administration.
15. Subjects who enrolled in another clinical trial and exposed to any investigational drug within 16 weeks of study enrollment.
16. Subjects who received blood infusion within 12 weeks, those who had blood drawn 400 mL or more within 12 weeks, 400 mL, or 200 mL or more within 4 weeks, or sampling of a component of the blood within 2 week of study drug administration.
17. Subjects who performed extreme exercises or exhausting labors (more than 1 hr/day or 5 day/week) within 2 weeks before hospitalization.
18. Any subject who, or whose partner, does not want to take highly reliable contraceptive measures until the end of the post-treatment examination.
19. Subjects who are inappropriate to participate in the study, as judged by the investigator or subinvestigator

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
PK Parameter Cmax, calculated from plasma E2020 concentration by a non-compartmental analysis, will be evaluated. | Up to 168 hrs after administration
PK Parameter AUC(0-168), calculated from plasma E2020 concentration by a non-compartmental analysis, will be evaluated. | Up to 168 hrs after administration

CONTACTS AND LOCATIONS:
Overall Officials: Hiroki Shimizu, Study Director — Eisai Co., Ltd.
Locations (1):
- Sumida-ku, Tokyo, Japan